CLINICAL TRIAL: NCT03370783
Title: Acute Neuroimmune Effects of Alcohol Using Free Water Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Mollie Monnig, Assistant Professor of Behavioral and Social Sciences, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1608001583; P20GM103645 (NIH)
Record Dates: First submitted 2017-12-07; First posted 2017-12-12 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ethanol — Moderate alcohol consumption

SUMMARY:
This study examines the effects of moderate alcohol intake on the brain, the immune system, and cognition.

DETAILED DESCRIPTION:
The study involves a within-subjects, pre/post design to assess the effects of a moderate dose of alcohol on immune biomarkers, neurobiological measures, and cognitive functioning. The study recruits healthy adults (ages 21-45) from the community to complete the experimental protocol. Participants complete magnetic resonance imaging scans, blood sample collection, and cognitive testing in the context of alcohol consumption.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-45 years
* Able to speak and read English at least at 8th grade level
* Moderate self-reported alcohol use in the past year
* Body mass index in normal to overweight range
* Right-handed

Exclusion Criteria:

* History of heavy drinking
* Currently seeking alcohol or drug treatment
* Chronic disease requiring use of medication
* Recent antibiotic or probiotic use
* Chronic daily use of NSAIDs
* Chronic GI disorder
* Use of illicit drugs
* Major psychiatric disorder or suicidality
* Fainting, weakness, infection, excessive bruising, or distress resulting from standard blood draw
* Safety contraindication for MRI scan
* Inability to abstain from use of tobacco products prior to or during study
* Inability to abstain from use of cannabis prior to or during study
* Pregnant, nursing, or may become pregnant

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Immune biomarkers | 1-3 hours after alcohol intake

CONTACTS AND LOCATIONS:
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT03370783/ICF_000.pdf